CLINICAL TRIAL: NCT03101228
Title: Medical and Physiological Benefits and Mechanisms of Reduced Sitting Without Meeting the Current Physical Activity Recommendations
Brief Title: Medical and Physiological Benefits of Reduced Sitting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Collaborators: UKK Institute (Other)
Responsible Party: Principal Investigator, Ilkka Heinonen, Principal Investigator, University of Turku
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: T91/2017
Record Dates: First submitted 2017-03-24; First posted 2017-04-05 (Actual); Last update posted 2020-04-08 (Actual); Status verified 2020-04

CONDITIONS: Metabolic Syndrome; Physical Activity; Insulin Resistance; Cardiovascular Diseases
Keywords: Physical Activity; Metabolic Syndrome; Insulin Sensitivity; Cardiovascular Risk Factor; Sedentary Lifestyle; Accelerometry
MeSH Terms: conditions — Metabolic Syndrome; Motor Activity; Insulin Resistance; Cardiovascular Diseases; Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: A parallel-group randomised controlled trial
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the intervention, masking of the participants is not possible. Analyzing of the obtained data will be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reduced sitting (Experimental): Objectively measured daily inactive time will be reduced by one hour compared to the baseline.
  Interventions: Behavioral: Reduced sitting
- Control (No Intervention): Subjects will be guided to maintain their normal sedentary behaviour and physical activity habits.

INTERVENTIONS:
Behavioral: Reduced sitting — Subjects are guided to limit their sitting time during the day for 1 hour/day, by adding light activity with the help of an activity monitor. Subjects are not encouraged to increase their moderate to vigorous physical activity levels.
  Arms: Reduced sitting

SUMMARY:
The most important objective of this randomized controlled trial in subjects with increased cardiovascular and metabolic risk factors is to investigate whether only reduced daily sitting improves human cardiovascular and metabolic health during a six-month intervention. It is hypothesized and expected that only reduced sitting, without formal physical activity or exercise training, affects favorably cardiovascular and metabolic health.

ELIGIBILITY:
Inclusion Criteria:

* Physically inactive (less than 120 minutes of moderate intensity exercise per week measured by the activity monitor during run-in)
* Sitting time ≥ 10 h /day (measured by the activity monitor during run-in)
* BMI 25-40
* Blood pressure < 160/100 mmHg
* Fasting plasma glucose < 7.0 mmol/l
* Fulfills the criteria of the metabolic syndrome according to Alberti et al 2009

Exclusion Criteria:

* History of a cardiac event
* Insulin or medically treated diabetes
* Any chronic disease or condition that could create a hazard to the subject safety, endanger the study procedures or interfere with the interpretation of study results
* Presence of ferromagnetic objects that would make MR imaging contraindicated
* Abundant use of alcohol
* Use of narcotics
* Smoking of tobacco or consuming snuff tobacco
* Diagnosed depressive or bipolar disorder
* Previous PET imaging or considerable exposure to radiation

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2017-04-25 (Actual); Primary Completion 2020-02-14 (Actual); Study Completion 2020-03-04 (Actual)

PRIMARY OUTCOMES:
The change in whole-body insulin sensitivity | The change from baseline to 6 months
  M-value during the hyperinsulinemic euglycemic clamp
The change in skeletal muscle insulin-stimulated glucose uptake | The change from baseline to 6 months
  Glucose uptake in the femoral muscles will be measured by positron emission tomography (PET) with [18F]-labelled fluoro-deoxy-glucose (FDG) tracer during hyperinsulinemic euglycemic clamp

SECONDARY OUTCOMES:
daily sitting hours | through study completion, an average of 6 months
  Accelerometry data will be collected during the whole intervention period by a triaxial hip-mounted accelerometer
daily hours spent physically active | through study completion, an average of 6 months
  Accelerometry data will be collected during the whole intervention period by a triaxial hip-mounted accelerometer
The change in liver adiposity | The change from baseline to 6 months
  Liver fat content will be assessed using magnetic resonance spectroscopy (MRS)
The change in maximal oxygen uptake | The change from baseline to 6 months
  Maximal oxygen uptake (VO2peak) will be determined by cycle ergometry with direct respiratory measurements. Exercise intensity will be started at 50 W and the intensity will be increased by 25 W at every two minutes until the criteria used to establish the VO2peak are met. The criteria used to establish the VO2peak are a plateau in VO2 despite of an increase in intensity and a respiratory quotient greater than 1.1. or volitional fatigue.
The change in body fat percentage | The change from baseline to 3 months
  Air displacement plethysmography (the Bod Pod system, COSMED, Inc., Concord, CA, USA) will be used to measure body composition (fat mass and fat free mass) with thoracic gas volume being predicted.
The change in body fat percentage | The change from baseline to 6 months
  Air displacement plethysmography (the Bod Pod system, COSMED, Inc., Concord, CA, USA) will be used to measure body composition (fat mass and fat free mass) with thoracic gas volume being predicted.
The change in plasma glucose | The change from baseline to 3 months
  Plasma glucose content will be measured from fasting venous blood samples using standard assays
The change in plasma glucose | The change from baseline to 6 months
  Plasma glucose content will be measured from fasting venous blood samples using standard assays
The change in HbA1c | The change from baseline to 3 months
  Glycated hemoglobin will be measured from fasting venous blood samples using standard assays
The change in HbA1c | The change from baseline to 6 months
  Glycated hemoglobin will be measured from fasting venous blood samples using standard assays

CONTACTS AND LOCATIONS:
Overall Officials: Juhani Knuuti, Professor, Study Chair — Turku PET Centre, Turku University Hospital
Locations (1):
- Turku PET Centre, Turku, Finland

IPD SHARING:
Plan to Share IPD: Undecided
IPD of the main outcome measures will be opened if possible.

REFERENCES:
- [Derived] Norha J, Sjoros T, Garthwaite T, Laine S, Laitinen K, Houttu N, Vaha-Ypya H, Sievanen H, Loyttyniemi E, Vasankari T, Knuuti J, Kalliokoski KK, Heinonen IHA. Secondary analysis of a randomised controlled trial on reducing sedentary behaviour and its effects on quality of life and wellbeing. Sci Rep. 2025 Oct 22;15(1):36861. doi: 10.1038/s41598-025-20836-7. PMID 41125692
- [Derived] Garthwaite T, Sjoros T, Laine S, Koivumaki M, Vaha-Ypya H, Norha J, Kallio P, Saarenhovi M, Loyttyniemi E, Sievanen H, Houttu N, Laitinen K, Kalliokoski KK, Vasankari T, Knuuti J, Heinonen I. Successfully Reducing Sitting Time Can Improve Metabolic Flexibility. Scand J Med Sci Sports. 2025 Aug;35(8):e70113. doi: 10.1111/sms.70113. PMID 40781908
- [Derived] Ylinen VP, Sjoros T, Laine S, Garthwaite T, Norha J, Vaha-Ypya H, Loyttyniemi E, Houttu N, Laitinen K, Kalliokoski KK, Sievanen H, Vasankari T, Knuuti J, Heinonen IH. Sedentary behavior reduction and blood lipids in adults with metabolic syndrome: a 6-month randomized controlled trial. Sci Rep. 2024 Oct 16;14(1):24241. doi: 10.1038/s41598-024-75579-8. PMID 39414998
- [Derived] Norha J, Sjoros T, Garthwaite T, Laine S, Verho T, Saunavaara V, Laitinen K, Houttu N, Hirvonen J, Vaha-Ypya H, Sievanen H, Loyttyniemi E, Vasankari T, Kalliokoski K, Heinonen I. Effects of reducing sedentary behaviour on back pain, paraspinal muscle insulin sensitivity and muscle fat fraction and their associations: a secondary analysis of a 6-month randomised controlled trial. BMJ Open. 2024 Sep 28;14(9):e084305. doi: 10.1136/bmjopen-2024-084305. PMID 39343453
- [Derived] Sjoros T, Norha J, Johansson R, Laine S, Garthwaite T, Vaha-Ypya H, Loyttyniemi E, Kalliokoski KK, Sievanen H, Vasankari T, Knuuti J, Heinonen IHA. Tiredness after work associates with less leisure-time physical activity. Sci Rep. 2024 Apr 4;14(1):7965. doi: 10.1038/s41598-024-58775-4. PMID 38575674
- [Derived] Sjoros T, Laine S, Garthwaite T, Vaha-Ypya H, Loyttyniemi E, Koivumaki M, Houttu N, Laitinen K, Kalliokoski KK, Sievanen H, Vasankari T, Knuuti J, Heinonen IHA. Reducing Sedentary Time and Whole-Body Insulin Sensitivity in Metabolic Syndrome: A 6-Month Randomized Controlled Trial. Med Sci Sports Exerc. 2023 Mar 1;55(3):342-353. doi: 10.1249/MSS.0000000000003054. Epub 2022 Oct 13. PMID 36251378
- [Derived] Norha J, Hautala AJ, Sjoros T, Laine S, Garthwaite T, Knuuti J, Loyttyniemi E, Vaha-Ypya H, Sievanen H, Vasankari T, Heinonen IHA. Standing time and daily proportion of sedentary time are associated with pain-related disability in a one month accelerometer measurement in adults with overweight or obesity. Scand J Pain. 2021 Sep 27;22(2):317-324. doi: 10.1515/sjpain-2021-0108. Print 2022 Apr 26. PMID 34582633
- [Derived] Sjoros T, Vaha-Ypya H, Laine S, Garthwaite T, Lahesmaa M, Laurila SM, Latva-Rasku A, Savolainen A, Miikkulainen A, Loyttyniemi E, Sievanen H, Kalliokoski KK, Knuuti J, Vasankari T, Heinonen IHA. Both sedentary time and physical activity are associated with cardiometabolic health in overweight adults in a 1 month accelerometer measurement. Sci Rep. 2020 Nov 25;10(1):20578. doi: 10.1038/s41598-020-77637-3. PMID 33239818